CLINICAL TRIAL: NCT00677742
Title: Impact of Pack Supply on Oral Contraception Continuation
Brief Title: The Impact of Pack Supply on Birth Control Pill Continuation
Acronym: SixPack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAC1723; 1 FPRPA0060250100
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Oral Contraception
Keywords: oral contraception; hormonal contraception; contraceptive behavior; patient compliance
MeSH Terms: conditions — Contraception Behavior; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): enhanced initial supply of oral contraception
  Interventions: Other: enhanced initial supply of oral contraception
- 2 (Active Comparator): conventional initial supply of oral contraception
  Interventions: Other: conventional initial supply of oral contraception

INTERVENTIONS:
Other: enhanced initial supply of oral contraception — 7 packs of pills, or 1 pack of pills and a prescription for 6 refills
  Arms: 1
Other: conventional initial supply of oral contraception — 3 packs of pills, or 1 pack of pills and a prescription for 2 refills
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether getting more packs of birth control pills leads to improved continuation, when compared with getting the traditional supply.

DETAILED DESCRIPTION:
Discontinuation of oral contraceptive use in the initial months is common; successful early continuation is predictive of long term continuation and prevention of unintended pregnancy. The conventional approach to initiation of hormonal contraceptives in publicly funded clinics across the United States is to give the patient a limited supply of OCs, or a prescription with a limited number of refills, and then have her return to the clinic for a refill. This approach requires the patient to make frequent visits to the clinic, a barrier to method continuation.

This randomized trial will evaluate a simple but potentially powerful change in family planning clinic practice, i.e., the effect of dispensing more versus fewer cycles of oral contraception (OC). The study will be carried out in an urban, publicly funded family planning clinic that serves a population that is poor, young and primarily Hispanic or AfricanAmerican. This population was targeted as its members are at increased risk of discontinuing contraception in the ﬁrst year of use.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaker
* age less than or equal to 35 years requesting OC as their primary method of contraception
* currently sexually active or anticipating sexual activity within the next 30 days

Exclusion Criteria:

* contraindications to oral contraceptives per clinic protocol (e.g., hypertension and pregnancy)
* currently using OCs (that is, current users requesting a routine refill)
* desiring pregnancy within the next 6 months
* leaving the clinic catchment area within 6 months
* previous participation in this study

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 700 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
oral contraception continuation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katharine O'Connell, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Family Planning Clinic, New York, New York, United States

REFERENCES:
- [Derived] White KO, Westhoff C. The effect of pack supply on oral contraceptive pill continuation: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):615-622. doi: 10.1097/AOG.0b013e3182289eab. PMID 21860291